CLINICAL TRIAL: NCT00359307
Title: Chemokine System Polymorphisms and Risk of Atherosclerosis (CAD)
Brief Title: Genetic Factors in Atherosclerosis
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000143; 00-I-0143
Record Dates: First submitted 2006-08-01; First posted 2006-08-02 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2013-03-21

CONDITIONS: Atherosclerosis
Keywords: Genetic; Longitudinal; Prospective; Epidemiology; Heart Attack
MeSH Terms: conditions — Atherosclerosis; Myocardial Infarction

SUMMARY:
The purpose of this study is to identify genes associated with certain risk factors for atherosclerosis (hardening of the arteries) and its consequences, such as development of coronary artery disease, heart attack, other blood vessel disease and stroke.

People enrolled in the Framingham Heart Study in Framingham, Massachusetts, are eligible to participate in this study. They will undergo a medical history, including review of their medical records and a family history; evaluation of memory and mood; breathing test and electrocardiogram (EKG); blood and urine tests, including blood sample collection for DNA (genetic) testing; evaluation of gait (walking), balance and hand grip strength; and hearing test. They will also fill out questionnaires on their eating habits and general health.

Any patients who may suffer a stroke during the study will be examined during their hospitalization and at 3, 6, 12, and 24 months after the stroke. This examination includes a neurological evaluation, assessment of ability to perform daily living tasks and, possibly, magnetic resonance imaging (MRI) of the brain, a test that uses a strong magnetic field and radio waves to produce pictures of the brain.

DETAILED DESCRIPTION:
We are studying the relationship between genetic variants of the human immune system and atherosclerosis through a collaboration with the Framingham Heart Study. Since atherosclerosis is a disease of chronic inflammation of the arterial vessel wall, genetic variants in molecules that are responsible for the migration of leukocytes are likely to explain some of the genetic diversity in the rate of heart disease and strokes. Therefore we are conducting a molecular epidemiology study of the genetics of atherosclerosis using materials and clinical data already collected by the Framingham Heart Study. The Heart Study is a prospective epidemiological study of the natural history of heart disease and stroke that has involved individuals residing in Framingham, Massachusetts since the 1950s. We will compare risks of individuals with particular genotypes for developing atherosclerosis and its sequelae, coronary artery disease, heart attack, peripheral vascular disease, and stroke. If correlations of genotype with risk of atherosclerosis can be found, then this will facilitate new treatments of this disease based on interference with particular components of the human immune system.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Free of acute and chronic diseases (especially GI disorders) as determined by medical history, physical examination and laboratory tests.
* Individuals may be taking antacids and/or laxative drugs but they must be discontinued 3 or more weeks before admission.
* Age 18-45 years (in order to minimize the effect of aging on nutrient absorption).
* BMI 18-25 kg/m(2) or greater than 35 kg/m(2).

EXCLUSION CRITERIA:

* History or clinical manifestation of:

  1. Current smoking
  2. Type 2 diabetes (according to the World Health Organization diagnostic criteria)
  3. Endocrine disorders, such as Cushing's disease, pituitary disorders, and hypo- and hyperthyroidism
  4. HIV infection (self-report), due to effects on weight and body composition of HIV and medications used to treat HIV
  5. Active tuberculosis (self-report)
  6. Pulmonary disorders, including physician diagnosed chronic obstructive pulmonary diseases and obstructive sleep apnea syndrome; only subjects with mild or exercise-induced asthma on no medications or on beta-adrenergic agonists only (such as albuterol) will be allowed to enter the study
  7. Cardiovascular diseases, including coronary heart disease, heart failure, arrhythmias, and peripheral artery disease
  8. Hypertension (according to the World Health Organization diagnostic criteria), treated or uncontrolled
  9. Gastrointestinal disease, including inflammatory bowel diseases (e.g. Crohn's disease and ulcerative colitis), malabsorption syndromes (e.g. celiac disease), gastric ulcer (active)
  10. Lactose intolerance
  11. Liver disease, including non-alcoholic fatty liver disease, AST or ALT greater than 1.5 x normal value, cirrhosis, active hepatitis B or C
  12. Renal disease, as defined by serum creatinine concentrations greater than 1.5 mg/dl and/or overt proteinuria
  13. Central nervous system disease, including previous history of cerebrovascular accidents, dementia, and neurodegenerative disorders
  14. Cancer requiring treatment in the past five years, except for non-melanoma skin cancers or cancers that have clearly been cured or, in the opinion of the investigator, carry an excellent prognosis
* Behavioral or psychiatric conditions that would be incompatible with a safe and successful participation in the study (such as major depression, schizophrenia and presence of psychotic symptoms)
* Taking weight loss drugs
* Use of any antibiotic or probiotic agents within the 2 months prior to the study
* Evidence of alcohol and/or drug abuse (more than 3 drinks per day and use of drugs, such as amphetamines, cocaine, heroin, or marijuana)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1888 (Actual)
Dates: Start 2000-06-08; Study Completion 2013-03-21

CONTACTS AND LOCATIONS:
Overall Officials: David H McDermott, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States